CLINICAL TRIAL: NCT06837831
Title: Efficacy of Mepilex Lite Dressings Combined with Indomethacin Suppositories in the Treatment of Anal Pain in Patients Undergoing Radiotherapy for Rectal Cancer: Protocol for a Randomized Controlled Trial
Brief Title: Efficacy of Mepilex Lite Dressings in Treating Anal Pain
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Qianfoshan Hospital (Other)
Responsible Party: Principal Investigator, Heli Shang, Associate Chief Nurse, Qianfoshan Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Zlflk2025
Record Dates: First submitted 2025-02-17; First posted 2025-02-20 (Actual); Last update posted 2025-02-25 (Actual); Status verified 2024-12

CONDITIONS: Rectal Cancer, Radiotherapy; Anal Pain
Keywords: Rectal cancer; mepilex lite dressings; indomethacin suppository; anal pain
MeSH Terms: conditions — Rectal Neoplasms | interventions — Control Groups

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control group (Other): Routine care
  Interventions: Other: Control group
- Experimental group (Experimental): mepilex lite dressings combined with indomethacin suppositories
  Interventions: Combination Product: Experimental group

INTERVENTIONS:
Other: Control group — Give routine nursing measures. Symptom management: Participants were informed that the damage to the anal canal mucosa caused by radiotherapy was mainly manifested as anal pain, and diarrhea could aggravate the symptoms of anal pain. Therefore, the patient should be instructed to monitor the symptoms of diarrhea and anal pain and give timely feedback; Dietary guidance: eat high-protein, high-vitamin, low-slag, low-fiber food, do not eat spicy and irritating food; Medication guidance: Follow the doctor's advice to take the drug orally on time and according to the amount, cooperate with the retention enema, etc., observe the effect of medication; Psychological guidance: strengthen nurse-patient communication, give psychological counseling, and rationally vent anxiety and other emotions. Perianal skin care: Wear loose cotton underwear to keep the perianal area clean and dry.
  Arms: Control group
Combination Product: Experimental group — After the patient emptied urine and feces before going to bed (21:00), the patient was assisted to take the kneeling lateral position, and the anal canal was cleaned with 0.9%Nacl soaked cotton swab, and was fully left to dry. After 30min, the anal pain was relieved. The operator fully exposed the patient's anus and part of the anal canal mucosal lesions with his left thumb and index finger, and applied a 6cm*6cm adhesive foam dressing on the injured mucosa with his right hand. With the help of a cotton swab, the patient was instructed to take a deep breath, send the foam dressing to 3cm of the anal canal, reveal 2cm, slowly release the left hand, withdraw the cotton swab at the same time the anus automatically retracted, which played a role in securing the dressing, and ask the patient to lie flat and rest, and take it out the next morning (06:00).
  Arms: Experimental group

SUMMARY:
BACKGROUND: Rectal cancer is a common gastrointestinal tumor, and low and intermediate rectal cancer accounts for 90% of rectal cancer. Radiotherapy is one of the important means of rectal cancer treatment, but the radiotoxicity induced by radiotherapy should not be neglected. As normal tissues around the target organ of radiotherapy, the anal canal is damaged by radiation and mucous membrane damage occurs, which is manifested as mucous membrane congestion, edema and ulceration, etc., and pain in the anal area occurs. With the accumulation of radiotherapy dose, the mucosal damage of the anal canal becomes more and more serious, and the anal pain of the patients is severe, which seriously affects the life quality of the patients. Therefore, the main objective of this study is to determine the effectiveness of mepilex lite dressings combined with indomethacin suppositories in the treatment of anal pain in patients undergoing radiotherapy for low and intermediate rectal cancer.

METHODS: The study protocol will be a single-blind randomized controlled trial. A randomized grouping method was used to divide the participants into an observation group (n=98) and a control group (n=98). The control group was given routine nursing measures, and the experimental group was given mepilex lite dressings for intra-anal insertion combined with indomethacin suppository for anal administration on the basis of routine nursing measures. The primary outcome indicator was anal pain score. Secondary outcome indicators were anxiety score, sleep quality score and comfort score. Assessments were made at baseline (anal pain NRS score ≥7 in patients undergoing radiotherapy for low to intermediate rectal cancer), day 1, day 7 and day 14 post-intervention. Statistical analyses will be performed using SPSS 25.0 and a significance level of p≤0.05 will be used for all tests.

DETAILED DESCRIPTION:
Outcome Measures:

1. Anal pain assessment: The degree of anal pain in patients was evaluated using the Numerical Rating Scale (NRS score), with 0-10 points representing different levels of pain. A score of 0 indicates no pain, 1-3 indicates mild pain, 4-6 indicates moderate pain, and 7-10 indicates severe pain. The higher the score, the more severe the pain. [22] For patients with middle and lower rectal cancer undergoing radiotherapy who experienced anal pain and had an NRS score of ≥7, evaluations were conducted on the first day, the seventh day, and the fourteenth day after intervention.
2. Anxiety assessment: The Self-Rating Anxiety Scale (SAS) was used to evaluate the degree of anxiety. The scale consists of 20 items, each scored from 1 to 4 points. The sum of the scores of all items is the total raw score. The SAS standard score is obtained by multiplying the total raw score by 1.25 and rounding to the nearest integer. The higher the score, the more severe the patient's anxiety.
3. Sleep quality assessment: The Pittsburgh Sleep Quality Index (PSQI) was used to evaluate the sleep quality and sleep disorders of the study participants. The PSQI consists of 19 self-rated items and 5 other-rated items.
4. Comfort assessment: The Chinese version of the General Comfort Questionnaire (GCQ) developed by American comfort care expert Kolcaba was adopted. It consists of four dimensions: physical, psychological and spiritual, sociocultural, and environmental, with a total of 28 items.

ELIGIBILITY:
Inclusion Criteria:

* (1) Patients with low and intermediate rectal cancer confirmed by pathological histologic diagnosis; (2) Patients who received radiotherapy; (3) Anal pain numerical rating scale (Numerical Rating Scale,NRS) ≥7 points; (4) Age ≥18 years; (5) Those who volunteered to participate in this study.

Exclusion Criteria:

1. Allergy, allergy to the drugs used in this study;
2. Mental illness, emotional instability or inability to express their feelings;
3. Combined serious cardiovascular and cerebrovascular diseases, digestive system diseases, blood system diseases and infectious diseases;
4. Previous history of pelvic radiotherapy;
5. Physical strength score (PS score) > 3 points -

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 196 (Estimated)
Dates: Start 2024-12-06 (Actual); Primary Completion 2026-12-06 (Estimated); Study Completion 2026-12-06 (Estimated)

PRIMARY OUTCOMES:
Assessment of anal pain | Patients with rectal pain and NRS score ≥7 were evaluated at baseline，Assessment was performed again on day 1, day 7, and day 14 after intervention
  A digital scoring method (NRS score) was used to evaluate the degree of anal pain of patients. 0-L0 scores were used to replace different degrees of pain. 0 scores meant no pain, 1-3 was classified as mild pain, 4-6 was classified as moderate pain, and 7-l0 was classified as severe pain

CONTACTS AND LOCATIONS:
Overall Officials: Heli Shang, undergraduate, Study Director — Shandong First Medical University
Locations (1):
- The First Affiliated Hospital of Shandong First Medical University, Jinan, Shandong, China

IPD SHARING:
Plan to Share IPD: Yes
Study Protocol
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: 1. The publication time of the study protocol and informed consent form shall be the time when the clinicaltrial approval is obtained.
  2. Statistical analysis plan and clinical study report will be published after the paper,about February 1, 2027.
  3. The above information is valid for 3 years after publication
Access Criteria: Everyone can access it at clinicaltrial or by emailing it directly at 15863788372@163.com.They have access to study protocols, statistical analyses, informed consent forms.